CLINICAL TRIAL: NCT04792736
Title: Prognostic Value of Lactates in Predicting Intensive Care Unit Mortality
Brief Title: Prognostic Value of Lactates in ICU
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of ICU department, Mongi Slim Hospital
Other Study IDs: Lactates ICU
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Mortality
Keywords: Lactates; Prognosis; intensive care units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Patients discharged alive from intensive care unit
  Interventions: Diagnostic Test: Blood lactate level
- non survivors: Patients who succumbed during their ICU stay
  Interventions: Diagnostic Test: Blood lactate level

INTERVENTIONS:
Diagnostic Test: Blood lactate level — Blood lactate level measured at admission H0, every 6 hours during the first 24 h and at H48

SUMMARY:
he aim of this prospective, analytic trial was to evaluate the accuracy of blood lactates levels in predicting mortality in ICU patients.

DETAILED DESCRIPTION:
In this study, conducted over o 12 months period, arterial blood lactates levels were measured in ICU patients at admission (H0), every 6 hours during the first day and and H48.

This trial included traumatic, medical and surgical patients requiring ICU stay for a predictive period > to 24 hours.

Blood lactates were evaluated as a prognostic parameter in predicting ICU mortality and compared to classic prognostic scores such as: SOFA score, IGS II and APACHE II.

The primary end point was ICU mortality.

ELIGIBILITY:
Inclusion Criteria:

* All adults admissions in ICU with a predicted length of stay > 24 hours

Exclusion Criteria:

* Patients who died during the first 24 hours after ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted in ICU after major trauma or surgery or for medical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | 28 days after ICU admission
  Mortality at Day 28

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - Mongi Slim University Hospital, La Marsa, Tunis Governorate
  - Mongi Slim Hospital, Tunis

IPD SHARING:
Plan to Share IPD: No